CLINICAL TRIAL: NCT04387734
Title: Effects and Mechanisms of Ocrevus on Ambulatory Functions in People With Relapsing Multiple Sclerosis
Brief Title: Effects of Ocrevus in Relapsing Multiple Sclerosis
Acronym: MOBILE-RMS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Multiple Sclerosis Center of Atlanta (Other)
Responsible Party: Principal Investigator, Feng Yang, PhD, Associate Professor, Georgia State University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RO-IIS-2019-20273
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Mobility; Fall risk; Balance; Multiple sclerosis; T2LV
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ocrevus (Experimental)
  Interventions: Drug: Ocrelizumab
- Other Disease Modifying Treatments (Active Comparator): Other Disease Modifying Treatments will consist of FDA-approved injectable and oral medications for multiple sclerosis.
  Interventions: Drug: Platform

INTERVENTIONS:
Drug: Ocrelizumab — Ocrevus will be administered following the FDA's regulations.
  Other Names: Ocrevus
  Arms: Ocrevus
Drug: Platform — The applications of the platform DMTs will follow the FDA-approved regulations.
  Other Names: Other injectable Disease Modification Treatments
  Arms: Other Disease Modifying Treatments

SUMMARY:
The purpose of this study is to test if people with relapsing multiple sclerosis (RMS) can improve ambulatory functions after one-year treatment with Ocrevus in comparison with other Disease Modifying Treatments (DMT). Sixty qualified individuals with RMS will be evenly assigned into two groups: Ocrevus and other DMT. Each group will receive the respective treatment following the FDA regulations over the one-year course. Their ambulatory functions will be assessed five times three months apart. In addition, they will receive brain MRI scans three times six months apart. Their ambulatory functions and MRI measurements will be compared between groups over time to fulfill the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written, informed consent and to be compliant with the schedule of protocol assessments;
2. Ages 18-65 years old at screening;
3. Clinically confirmed active, relapsing forms of MS (RMS) based on the revised McDonald criteria;
4. Can walk at least 25 feet independently with or without assistive device at screening (or the Expanded Disability Status Scale between 1 and 6.5);
5. Can stand independently for at least 30 seconds;
6. Not pregnant at screening and throughout the study;
7. No other neurological conditions and recent musculoskeletal injuries;
8. Can read and understand English;
9. No significant cognitive impairment.

Exclusion Criteria:

1. History of other types of MS at screening such as, primary-progressive MS);
2. Inability to complete an MRI (contraindications for MRI include but are not limited to claustrophobia, body mass greater than 140 kg, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks before the time of the intended MRI, etc);
3. Patients with an active hepatitis B virus (HBV) infection;
4. Have a life-threatening allergic reaction to ocrelizumab or any of its ingredients in the past;
5. Hypersensitive to any of the ingredients of ocrelizumab;
6. Do not understand English.

   Exclusions related to general health
7. Pregnancy or lactation;
8. Have any other known neurological diseases which may mimic MS including but not limited to: Neuromyelitis optica, Lyme disease, untreated vitamin B12 deficiency, neurosarcoidosis, and cerebrovascular disorders;
9. Suffering from coexisting psychiatric disorders, neurological disorders, or severe medical illness;
10. Current severe depression and/or suicidal ideation;
11. Significant cognitive impairment (Montreal Cognitive Assessment score < 24);
12. New onset, unstable orthopedic comorbid diagnoses (within 3 months and uncontrolled);
13. History or currently active primary or secondary immunodeficiency;
14. Receipt of a live vaccine within 6 weeks prior to baseline;
15. Skin is allergic to transparent double-side tapes;
16. Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study;
17. History or currently active primary or secondary immunodeficiency;
18. Lack of peripheral venous access;
19. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies;
20. Significant or uncontrolled somatic disease or any other significant disease that may preclude patient from participating in the study;
21. Congestive heart failure (NYHA III or IV functional severity);
22. Known active bacterial, viral, fungal, mycobacterial infection or other infection, excluding fungal infection of nail beds;
23. Infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit;
24. History or known presence of recurrent or chronic infection (e.g., hepatitis B or C, HIV, syphilis, tuberculosis);
25. History of progressive multifocal leukoencephalopathy (PML);
26. History of malignancy, including solid tumors and hematological malignancies, except basal cell carcinoma, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix of the uterus that have been previously completely excised with documented, clear margins;
27. History of alcohol or drug abuse within 24 weeks prior to baseline;
28. History or laboratory evidence of coagulation disorders;

    Exclusions related to medications
29. Receipt of a live vaccine within 6 weeks prior to baseline;
30. Treatment with any investigational agent within 24 weeks of screening (Visit 1) or five half-lives of the investigational drug (whichever is longer);
31. Contraindications to or intolerance of oral or intravenous corticosteroids, including methylprednisolone administered intravenous, according to the country label, including:

    1. Psychosis not yet controlled by a treatment;
    2. Hypersensitivity to any of the constituents;
32. Treatment with dalfamipridine (Ampyra®) unless on stable dose for ≥ 30 days prior to screening. Patients should remain on stable doses throughout the 52-week treatment period;
33. Previous treatment with B-cell targeted therapies (i.e. rituximab, ocrelizumab, atacicept, belimumab or ofatumumab);
34. Systemic corticosteroid therapy within 4 weeks prior to screening;
35. Any previous treatment with alemtuzumab (Campath), anti-CD4, cladribine, mitoxantrone, daclizumab, BG12, teriflunomide, laquinimod, total body irradiation or bone marrow transplantation;
36. Treatment with cyclophosphamide, azathioprine, mycophenolate mofetil (MMF), cyclosporine, methotrexate, or natalizumab within 24 months prior to screening;
37. Treatment with intravenous immunoglobulin within 12 weeks prior to baseline.

    Exclusions related to motor function
38. Cannot walk at least 25 feet and stand at least 30 seconds independently;
39. Weak or blind vision may impair their ability of walking;

    Exclusions related to musculoskeletal, cardiovascular, and orthopedic condition
40. Broken bones as an adult in the past year;
41. Have received neurological treatment, such as Botox, in the past six months;
42. Heart attack, angioplasty, or coronary artery bypass graft in the past six months;
43. Congestive heart failure (NYHA III or IV functional severity);
44. Surgery on back, hip, shoulder, or total joint replacement of hip or knee joint less than two years ago;
45. Respiratory conditions (lung cancer, bronchitis, emphysema, asthma, shortness of breath) not under regular medical care or the patient is medically unstable.

    Exclusions related to laboratory findings
46. Positive serum β hCG measured at screening;
47. Positive screening tests for hepatitis B (hepatitis B surface antigen [HBsAg] positive, or positive hepatitis B core antibody [total HBcAb] confirmed by a positive viral deoxyribonucleic acid [DNA] polymerase chain reaction [PCR]) or hepatitis C (HepCAb);
48. Positive rapid plasma reagin (RPR);
49. CD4 count < 300/μL;
50. AST/SGOT or ALT/SGPT ≥ 2.0 Upper Limit of Normal (ULN);
51. Platelet count <100,000/μL (<100 x 109/L);
52. Levels of serum IgG <5.65 g/L;
53. Levels of serum IgM < 0.55 g/L;
54. Total neutrophil count <1.5 x 103/μL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Stability | 12 months
  To quantify dynamic balance of participants during level walking.

SECONDARY OUTCOMES:
Gait speed | 12 months
  To quantify the distance covered per second.
Step length | 12 months
  The length of the step.
Step width | 12 months
  The width of the step.
Step time | 12 months
  Time elapsed between heel-strike of the contralateral foot and the successive heel-strike of the ipsilateral foot
Cadence | 12 months
  To quantify the number of steps taken within one minute
Stability index | 12 months
  Sway index is to characterize the static postural control associated with three sensory systems in people with multiple sclerosis.
Swing index | 12 months
  Swing index is another matrix measuring static balance.
Lower limb muscle strength | 12 months
  The maximum voluntary muscle strength at bilateral knee and ankle joints.
Lower limb muscle activity | 12 months
  The electrical activity of leg muscles during level walking
Multiple Sclerosis Functional Composite | 12 months
  The assessment of the disability status based on lower extremity function, upper extremity function, and cognitive function.
Expanded Disability Status Scale | 12 months
  Another assessment of the level of disability in people with multiple sclerosis. The Expanded Disability Status Scale score ranges from 0 to 10 (in increments of 0.5). A smaller score indicates a lower level of disability.
Total cerebral T2 lesion volume | 12 months
  T2-weighted lesion volume has been used as a measure of disease progression in multiple sclerosis.
Prospective falls | 12 months
  The number of fall incidences occurred in everyday living, and the details of each fall (if any), including the date, environment, and possible causes will be recorded using a falls-questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yang, PhD, Principal Investigator — Georgia State University
Locations (2):
- United States (2):
  - Georgia State University, Atlanta, Georgia
  - Multiple Sclerosis Center of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No